CLINICAL TRIAL: NCT02317042
Title: The Evaluation of the Sleep-Breathing Treatment Algorithm: AutoEPAP iVAPS
Brief Title: Juno Perth Clinical Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Phase II not initiated for commercial reasons (no safety related issues)
Sponsor: ResMed (Industry)
Collaborators: Sir Charles Gairdner Hospital (Other); The University of Western Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MA250814
Record Dates: First submitted 2014-12-08; First posted 2014-12-15 (Estimated); Results first posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Respiratory Insufficiency; Obesity Hypoventilation Syndrome; Chronic Obstructive Pulmonary Disease (COPD); Neuromuscular Disease; Upper Airway Obstruction
MeSH Terms: conditions — Respiratory Insufficiency; Obesity Hypoventilation Syndrome; Pulmonary Disease, Chronic Obstructive; Neuromuscular Diseases; Airway Obstruction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard ST Mode (Active Comparator): Participants underwent the first PSG study (Titration Night 1) on ST Mode ( prior to going on AutoEPAP iVAPS or Fixed EPAP iVAPS) whilst receiving their standard NIV therapy through the clinical trial device "Juno". During this mode the participant's current NIV settings were reviewed and re-titrated to deliver optimal therapy.
  Interventions: Device: Juno
- AutoEPAP iVAPS (Experimental): Participants underwent a PSG study on the AutoEPAP iVAPS mode on either Night 2 or Night 3 according to their computer generated randomisation.
  Participants were randomised (1:1) according to a computer-generated randomised list (Microsoft Excel 2010) to receive 'AutoEPAP iVAPS' or 'FixedEPAP iVAPS' therapy mode first.
  Interventions: Device: Juno
- Fixed EPAP iVAPS (Active Comparator): Participants underwent a PSG study on the Fixed EPAP iVAPS mode on either Night 2 or Night 3 according to their computer generated randomisation.
  Participants were randomised (1:1) according to a computer-generated randomised list (Microsoft Excel 2010) to receive 'AutoEPAP iVAPS' or 'FixedEPAP iVAPS' therapy mode first.
  Interventions: Device: Juno

INTERVENTIONS:
Device: Juno — Juno device set to ST mode with participant's current therapy settings.
  Other Names: ResMed "Juno" Device
  Arms: Standard ST Mode
Device: Juno — Juno device set to AutoEPAP iVAPS mode.
  Other Names: ResMed "Juno" Device
  Arms: AutoEPAP iVAPS
Device: Juno — Juno device set to Fixed EPAP iVAPS mode.
  Other Names: ResMed "Juno" Device
  Arms: Fixed EPAP iVAPS

SUMMARY:
This study is to evaluate the efficacy of a new therapy (Automatic Expiratory Positive Airway Pressure with intelligent Volume Assured Pressure Support (AutoEPAP iVAPS)) designed to treat respiratory insufficiency, respiratory failure and/or nocturnal hypoventilation with upper airway obstruction. The study will be performed in two phases: In a sleep unit and in the home environment. The new therapy will be compared against two existing ventilator therapies: "Spontaneous Timed (ST) mode" and "Intelligent Volume Assured Pressure Support (iVAPS)".

DETAILED DESCRIPTION:
Phase I: AutoEPAP iVAPS will be compared against two existing ventilator therapies: "Spontaneous Timed (ST) mode" and "Intelligent Volume Assured Pressure Support (Fixed EPAP iVAPS)" in current NIV users with respiratory insufficiency and /or respiratory failure due to Chronic Obstructive Pulmonary Disease (COPD),Obesity Hypoventilation Syndrome (OHS) or Neuromuscular Disease (NMD). Patients will spend a total of 3 nights in the sleep laboratory in the three modes described above. The apnoea-hypopnoea index will be the primary outcome measure.

Phase II: AutoEPAP iVAPS will be compared to ST mode over a period of 7 nights in the patients' home. The mean EPAP setting of each device will be the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria

* Subject has ability to provide written informed consent
* Subject aged ≥18 years old
* Subject has a diagnosis of COPD, OHS or NMD with sleep hypoventilation (historical PtCO2 increase overnight ≥ 10mmHg) and/or daytime hypercapnia (>45 mmHg)
* Subject is currently using non-invasive ventilation for ≥ 3 months
* Subject with an AHI ≥ 5 hr. (as documented in diagnostic or pressure determination sleep study report)

Exclusion Criteria

* Subjects not compliant on NIV (ie. < 4 hr/night)
* Subjects with severe asthma
* Subjects who are pregnant
* Subjects on oxygen therapy (ie. >4 L/min)
* Subjects with a tracheostomy
* Subjects who are acutely ill, medically complicated or who are medically unstable
* Subjects in whom PAP therapy is otherwise medically contraindicated
* Subjects who have had surgery of the upper airway, nose, sinus, or middle ear within the previous 90 days
* Subjects with untreated, non-OSA sleep disorders, including but not limited to; insomnia, periodic limb movement syndrome, or restless legs syndrome.
* Subjects who require ventilatory support during wakefulness
* Subjects with the following pre-existing conditions: severe bullous lung disease, recurrent pneumothorax or pneumomediastinum, low blood pressure, cerebrospinal fluid leak, recent cranial surgery or trauma.
* Subjects with severe developmental delay and who will not be able to follow tasks as instructed in the protocol.
* Subjects who the investigator believes are unsuitable for inclusion because either:

  * they do not comprehend English
  * they are unable or unwilling to provide written informed consent
  * they are physically unable to comply with the protocol
  * they are unsuitable to participate in the trial for any other reason in the opinion of the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-05-29 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Sir Charles Gairdner Hospital, Perth, Western Australia
  - University of Western Australia, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: An overnight PSG retitration was performed by experienced sleep technologists to ensure current EPAP & other device settings were optimal. Titration took place with the device in ST mode with the patient's usual therapy setup. If the device settings were not optimal or if other problems such as patient-device dysynchrony, then the ventilator settings were adjusted by the sleep technologist based on current guidelines. Retitration studies were reviewed by at least 2 experienced sleep physicians.
Groups:
- Standard ST Mode -> AutoEPAP iVAPS -> Fixed EPAP iVAPS: Night 1 Participants underwent the first PSG study on ST Mode receiving their standard NIV therapy through the clinical trial device "Juno". During this mode the participant's current NIV settings were reviewed and re-titrated to deliver optimal therapy.
  Night 2 Participants underwent a PSG study on the AutoEPAP iVAPS mode Night 3 Participants underwent a PSG study on the Fixed EPAP iVAPS mode
- Standard ST Mode -> FixedEPAP iVAPS -> AutoEPAP iVAPS Mode: Night 1 Participants underwent the first PSG study on ST Mode receiving their standard NIV therapy through the clinical trial device "Juno". During this mode the participant's current NIV settings were reviewed and re-titrated to deliver optimal therapy.
  Night 2 Participants underwent a PSG study on the FixedEPAP iVAPS mode Night 3 Participants underwent a PSG study on the AutoEPAP iVAPS mode
Period: Overall Study
Arm/Group | Standard ST Mode -> AutoEPAP iVAPS -> Fixed EPAP iVAPS | Standard ST Mode -> FixedEPAP iVAPS -> AutoEPAP iVAPS Mode
Started (Cross over design. 11/25 started with AutoEPAP and 14/25 started with FixedEPAP) | 11 | 14
Completed | 11 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Participant Baseline: Participant's meeting the eligibility criteria had their baseline information collected at their Visit 1.
Arm/Group | Participant Baseline
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Region of Enrollment [Number; unit: participants]
  Australia | 25

OUTCOME MEASURES:

1. Primary Outcome: Apnoea-Hypopnoea Index (AHI)
Description: The number of apneas and hypopnoeas per hour of sleep measured using AutoEPAP iVAPS versus Fixed EPAP iVAPS
Time Frame: 1 night
Population: Participants included in the study were those with a documented diagnosis of respiratory insufficiency and /or respiratory failure due to Chronic Obstructive Pulmonary Disease (COPD), Obesity Hypoventilation Syndrome (OHS) and Neuromuscular Disease (NMD).
Measure: Mean (Standard Deviation); unit: events/hour
Groups:
- Standard ST Mode: Participants underwent the first PSG study (Titration Night 1) on ST Mode whilst receiving their standard NIV therapy through the clinical trial device "Juno". During this mode the participant's current NIV settings were reviewed and re-titrated to deliver optimal therapy.
- FixedEPAP iVAPS: Participants underwent a PSG study on the Fixed EPAP iVAPS mode on either Night 2 or Night 3 according to their computer generated randomisation.
  Participants were randomised (1:1) according to a computer-generated randomised list (Microsoft Excel 2010) to receive 'AutoEPAP iVAPS' or 'FixedEPAP iVAPS' therapy mode first.
Arm/Group | Standard ST Mode | AutoEPAP iVAPS | FixedEPAP iVAPS
Number analyzed (Participants) | 25 | 25 | 25
events/hour | 3.87 (6.19) | 3.57 (3.76) | 4.09 (5.54)

2. Secondary Outcome: Oxygen Desaturation Index
Description: Number of oxygen desaturations per hour of sleep
Time Frame: 1 night
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | Standard ST Mode | AutoEPAP iVAPS | FixedEPAP iVAPS
Number analyzed (Participants) | 25 | 25 | 25
events/hour | 5.06 (6.18) | 4.45 (4.15) | 5.70 (8.96)

3. Secondary Outcome: Mean Oxygen Saturation
Description: Mean oxygen saturation recorded in the total sleep time
Time Frame: 1 night
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Standard ST Mode | AutoEPAP iVAPS | FixedEPAP iVAPS
Number analyzed (Participants) | 25 | 25 | 25
percentage of oxygen saturation | 93.99 (1.97) | 94.01 (1.89) | 94.33 (2.12)

4. Secondary Outcome: Time Spent Below 90% Oxygen Saturation
Description: Time in minutes that the oxygen saturation was below 90%
Time Frame: 1 night
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Standard ST Mode | AutoEPAP iVAPS | FixedEPAP iVAPS
Number analyzed (Participants) | 25 | 25 | 25
Minutes | 37.26 (78.18) | 37.03 (87.75) | 34.31 (100.25)

5. Secondary Outcome: Mean Transcutaneous Carbon Dioxide (PtcCo2)
Description: Transcutaneous Carbon Dioxide measurement (TcCO2)
Time Frame: 1 night
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Standard ST Mode | AutoEPAP iVAPS | FixedEPAP iVAPS
Number analyzed (Participants) | 24 | 24 | 24
mmHg | 45.73 (6.10) | 47.44 (5.04) | 46.78 (6.10)

6. Secondary Outcome: Sleep Duration
Description: Time spent asleep
Time Frame: 1 Night
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Standard ST Mode | AutoEPAP iVAPS | FixedEPAP iVAPS
Number analyzed (Participants) | 25 | 25 | 25
Minutes | 333.4 (86.06) | 331.7 (109.08) | 340.9 (110.43)

7. Secondary Outcome: Sleep Efficacy
Description: Sleep time divided by total time available for sleep
Time Frame: 1 Night
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of total recorded time
Arm/Group | Standard ST Mode | AutoEPAP iVAPS | FixedEPAP iVAPS
Number analyzed (Participants) | 25 | 25 | 25
percentage of total recorded time | 64 (15) | 66 (15) | 66 (18)

8. Secondary Outcome: Sleep Latency-Wake After Sleep Onset Time
Description: Time awake in minutes after initial sleep onset
Time Frame: 1 Night
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Standard ST Mode | AutoEPAP iVAPS | FixedEPAP iVAPS
Number analyzed (Participants) | 25 | 25 | 25
Minutes | 22.56 (17.41) | 29.98 (43.19) | 28.12 (29.98)

9. Secondary Outcome: Total Sleep Time Spent in Each Sleep Stage
Description: Percentage of total sleep time spent in each sleep stage (ie. N1, N2, N3 and REM)
Time Frame: 1 Night
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Standard ST Mode | AutoEPAP iVAPS | FixedEPAP iVAPS
Number analyzed (Participants) | 25 | 25 | 25
Minutes
  Time spent in N1 Sleep | 75.68 (33.88) | 76.62 (45.18) | 82.08 (46.31)
  Time spent in N2 Sleep | 186.9 (67.14) | 172.3 (74.08) | 174.9 (85.09)
  Time spent in N3 Sleep | 27.36 (26.43) | 37.38 (31.26) | 29.98 (24.73)
  Time spent in REM Sleep | 44.04 (26.36) | 45.30 (24.99) | 54.00 (44.10)

10. Secondary Outcome: Number of Respiratory Event Related Arousals/ Hour
Description: Total number of respiratory event related arousals/hr over the entire sleep period
Time Frame: 1 Night
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: arousals/hr
Arm/Group | Standard ST Mode | AutoEPAP iVAPS | FixedEPAP iVAPS
Number analyzed (Participants) | 25 | 25 | 25
arousals/hr | 5.17 (5.85) | 5.67 (4.14) | 6.54 (7.69)

11. Secondary Outcome: Number of Spontaneous Arousals/Hour
Description: Number of spontaneous arousals/hr occurring over the entire total sleep time
Time Frame: 1 Night
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: arousals/hr
Arm/Group | Standard ST Mode | AutoEPAP iVAPS | FixedEPAP iVAPS
Number analyzed (Participants) | 25 | 25 | 25
arousals/hr | 31.41 (21.09) | 29.21 (18.16) | 31.92 (23.67)

ADVERSE EVENTS:
Groups:
- Standard ST Mode: Standard ST mode.
- AutoEPAP iVAPS: AutoEPAP iVAPS.
- FixedEPAP iVAPS: FixedEPAP iVAPS.
Arm/Group | Standard ST Mode | AutoEPAP iVAPS | FixedEPAP iVAPS
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/25 | 0/25
Other Adverse Events (participants affected / at risk) | 4/25 | 2/25 | 2/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard ST Mode (N=25) | AutoEPAP iVAPS (N=25) | FixedEPAP iVAPS (N=25)
Multiple Falls (General disorders) | 0 (0) | 1 (2) | 0 (0) — Subject admitted to hospital following multiple falls which occurred after Titration Night 1. A rib fracture as a result of the SAE was noted at a later date. SAE and secondary event not related to study device or disease targeted by the trial.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard ST Mode (N=25) | AutoEPAP iVAPS (N=25) | FixedEPAP iVAPS (N=25)
Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1) | 0 (0)
AEROPHAGIA (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
SORE BACK (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
SKIN ABRASION TO CHIN (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
MILD CHEST INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has the right to

* review
* provide comments (site is not bound to follow them)
* request delay of publication for no more than 120 days to allow for securing of IP
* request the removal of specified confidential information

within 40 days of the proposed publication being released to those not bound by confidentiality obligations.